CLINICAL TRIAL: NCT01117077
Title: The Immune Tolerance Mechanism Induced by IL-17-producing Regulatory T Cells in the Orthotopic Liver Transplant Recipients With Aspergillosis
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Shanghai First People's Hospital, Shanghai First People's Hospital
Other Study IDs: 10ZR1423900
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Last update posted 2010-05-05 (Estimated); Status verified 2010-05

CONDITIONS: Liver Transplantation; Aspergillus; Interleukin-17; Treg Cell; Immune Tolerance
Keywords: liver transplantation; aspergillus infection; interleukin-17; Treg cell; immune tolerance
MeSH Terms: conditions — Aspergillosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Infection accounted for the first cause of death in patients after liver transplantation, and 2 / 3 of the cause of death was fungal infections. The investigators group early found that T cell subsets playing a role of inducing immune tolerance were significantly increased in vivo of liver transplantation patients with aspergillus infection, which may be a kind of Treg cells expressing IL-17. To explore the immune tolerance mechanism induced by the immune balance cells is important to liver transplantation patients for improving efficacy and reducing the mortality. Therefore, the investigators are going to get the blood sample and liver tissue of the liver transplantation patients before and after treatment of aspergillus infection, flow cytometry analysis of blood T cell subsets, Cytometric Bead Array to detect changes in blood cytokines, laser capture microdissection to obtain liver biopsies of inflammatory cells in portal area and further for analysis of T cell subsets and protein. And the investigators are also to investigate the characteristics of CCR6 + CD4 + FOXP3 + Treg cell clones secreting IL-17 and the capacity of which suppressing conventional T cell proliferation. This study may find new methods, such as certain types of T cell subsets or cytokines for the treatment of liver transplant patients, which not only to anti-rejection but also to reduce fungal infection.

ELIGIBILITY:
Inclusion Criteria:

Liver transplantation patients

Exclusion Criteria:

Psychopath

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: liver transplantation patients with aspergillus infection or without aspergillus infection
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-05